CLINICAL TRIAL: NCT02606240
Title: Extracorporeal CO2 Removal (ECCO2R) With a Renal Replacement Platform (PRISMALUNG) to Enhance Lung Protective Ventilation in Patients With Mild to Moderate Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Low-Flow CO2 Removal for Mild to Moderate ARDS With PRISMALUNG
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Centre Hospitalier Universitaire, Amiens (Other); Centre Hospitalier Universitaire de Besancon (Other); University Hospital, Clermont-Ferrand (Other); University Hospital, Montpellier (Other)
Responsible Party: Principal Investigator, Alain COMBES, Professor of Intensive Care Medicine, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: PSL-AC-11-11-15
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mild to Moderate ARDS on PRISMALUNG: Extracorporeal CO2 removal (ECCO2R) with the PRISMALUNG device in patients with mild to moderate Acute Respiratory Distress Syndrome (ARDS).
  Interventions: Device: CO2 removal with PRISMALUNG in ARDS

INTERVENTIONS:
Device: CO2 removal with PRISMALUNG in ARDS — Observational study of patients with mild to moderate Acute Respiratory Distress Syndrome (ARDS) submitted to Extracorporeal CO2 removal (ECCO2R) with the PRISMALUNG device to allow ultraprotective mechanical ventilation with tidal volume reduction (from 6 to 4 ml/kg, predicted body weight) and plateau pressure reduction from 28-30 to 23-25 cmH2O.

SUMMARY:
This pilot observational study will assess changes in pH /PaO2 /PaCO2, Respiratory Rate and device CO2 clearance in the first 24 hours of Extracorporeal CO2 removal (ECCO2R) following tidal volume (Vt), and plateau pressure reduction in patients with mild to moderate ARDS.

DETAILED DESCRIPTION:
Extracorporeal CO2 removal (ECCO2R) with a low-flow CO2 removal device (Prismalung, Gambro-Baxter) integrated on the Prismaflex platform (Gambro-Baxter) allows tidal volume (Vt) and plateau pressure reduction in patients with mild to moderate ARDS. This pilot observational study will assess changes in pH /PaO2 /PaCO2, Respiratory Rate and device CO2 clearance in the first 24 hours of ECCO2R following Vt and plateau pressure reduction in patients with mild to moderate ARDS. Safety variables during treatment will also be analyzed. A series of 20 consecutive patients will be included in this observational study.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation with expected duration of >24 hours
* Mild to moderate Acute Respiratory Distress Syndrome (ARDS) according to the Berlin definition: 100 mmHg <PaO2/FiO2 <300 mmHg, with PEEP > 5 cmH2O

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Severe hypoxemia with PaO2/FiO2 <100 mmHg
* Body mass index > 40 kg/m2
* Decompensated heart insufficiency or acute coronary syndrome
* Severe Chronic obstructive pulmonary disease (COPD)
* Major respiratory acidosis with PaCO2 >60 mmHg
* Acute brain injury
* Severe liver insufficiency (Child-Pugh scores >7) or fulminant hepatic failure
* Heparin-induced thrombocytopenia
* Contraindication for systemic anticoagulation
* Patient moribund, decision to limit therapeutic interventions
* Catheter access to femoral vein or jugular vein impossible
* Pneumothorax
* Platelet <50 G/L
* Lacking consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild to Moderate ARDS according to the Berlin definition of ARDS
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieved a tidal volume (Vt) reduction to 4 mL/kg while maintaining pH and PaCO2 to ± 20% of baseline values obtained at Vt of 6 mL/kg. | 24 hours
  Number of participants who achieved a tidal volume (Vt) reduction to 4 mL/kg while maintaining pH and PaCO2 to ± 20% of baseline values obtained at Vt of 6 mL/kg.

SECONDARY OUTCOMES:
Assessment of changes in Vt | 24 hours
  Assessment of changes in Vt
Assessment of changes in Plateau Pressure | 24 hours
  Assessment of changes in Plateau Pressure
Assessment of changes in respiratory rate | 24 hours
  Assessment of changes in respiratory rate
Assessment of changes in Positive End-Expiratory Pressure, PEEP | 24 hours
  Assessment of changes in Positive End-Expiratory Pressure, PEEP
Change in vasopressor use | 24 hours
  Epineprine and norepinephine dose, mcg/kg/min
Evaluation of lung recruitment/derecruitment | 24 hours
  With lung echography. Ccording to the method described by Bouhemad et al, Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7
Lifetime of the extracorporeal circulation | 7 days
  In hours
Number of participants with adverse events directly related to ECCO2R | 7 days
  Adverse events directly related to ECCO2R are hemolysis (serum free hemoglobin >500 mg/L), infection at the cannulation site, Hemorrhage at the cannulation site, air entry in the circuit.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU AMIENS, Département Anesthésie Réanimation, Amiens
  - CHU Besançon, Réanimation, Besançon
  - CHU CLERMONT FERRAND, Département Anesthésie Réanimation, Clermont-Ferrand
  - CHU MONTPELLIER, Département Anesthésie Réanimation, Montpellier
  - Hopital Pitié Salpetriere, Reanimation Medicale, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schmidt M, Jaber S, Zogheib E, Godet T, Capellier G, Combes A. Feasibility and safety of low-flow extracorporeal CO2 removal managed with a renal replacement platform to enhance lung-protective ventilation of patients with mild-to-moderate ARDS. Crit Care. 2018 May 10;22(1):122. doi: 10.1186/s13054-018-2038-5. PMID 29743094